CLINICAL TRIAL: NCT04761406
Title: Efficacy of a Microalgae Extract PhaeoSOL on Optimizing the Benefits of Healthy, Overweight and Moderately Obese Women Participating in an Exercise and Weight Management Program.
Brief Title: Microalgae Extract Phaeosol Combined to Exercise in Healthy Overweight Women : Efficacy on Body Weight Management
Acronym: PHAEOSOL-ONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microphyt (Industry)
Collaborators: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB2020-1443
Record Dates: First submitted 2021-02-08; First posted 2021-02-18 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Overweight and Obesity; Body Weight Changes; Healthy Lifestyle; Exercise; Dietary Supplement
Keywords: Fucoxanthin; Weight management; Microalgae; Exercise; Overweight
MeSH Terms: conditions — Overweight; Obesity; Body Weight Changes; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, double-blind, parallel arm intervention trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phaeosol group (Experimental): Daily supplementation of Phaeosol softgel capsule (218mg/d), active ingredients of Microphyt. Each randomized subject will consume 1 softgel capsule (before breakfast) per day during 12 weeks
  Interventions: Dietary Supplement: Phaeosol group
- Placebo group (Placebo Comparator): Daily supplementation of placebo softgel capsule (218mg/d of 100% sunflower oil) with the same appearance and packaging than experimental product. Each randomized subject will consume 1 softgel capsule (before breakfast) per day during 12 weeks
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Phaeosol group — In a double blind, randomized manner, 40 pre-menopausal females will ingest one of the following for 12 weeks:
  Treatment 1 -Placebo (218 mg/d of 100% sunflower Oil) Treatment 2 - PhaeoSOL (218 mg/d)
  Supplements will be prepared in softgel capsules for double blind administration by the sponsor.
  Arms: Phaeosol group
Dietary Supplement: Placebo group — In a double blind, randomized manner, 40 pre-menopausal females will ingest one of the following for 12 weeks:
  Treatment 1 -Placebo (218 mg/d of 100% sunflower Oil) Treatment 2 - PhaeoSOL (218 mg/d)
  Supplements will be prepared in softgel capsules for double blind administration by the sponsor.
  Arms: Placebo group

SUMMARY:
PhaoeSOL (Microphyt, Baillargues, France) is a microalgae-based nutritional ingredient developed with a patented production process that has New Dietary Ingredient (NDI) status from the FDA (#1120). It is an extract of the microalgae Phaeodactylum tricornutum standardized to 2.0% Fucoxanthin (FX) content by adding a food grade medium-chain triglyceride (MCT)-oil and a tocopherol-rich (Vitamin E) extract (0.5 % w:w). PhaeoSOL is intended for use as a source of the naturally occurring carotenoid, fucoxanthin, in food supplement products for the general population at levels not to exceed 437 mg/person/day for a maximal duration of 30 days of PhaeoSOL (equivalent to 10 mg fucoxanthin/person/day). Prior studies suggest that marine algae and Fucoxanthinol may have anti-obesity, lipid lowering, and glucose management enhancing properties. The purpose of this proof of concept pilot study is to examine whether dietary supplementation of PhaoeSOL enhances the benefits of women participating in an exercise and weight management program.

DETAILED DESCRIPTION:
All participants will participate in a supervised exercise training 3 days per week at the HCRF consisting of a 5-min warm-up, light stretching, resistance training (3 sets of 10 repetitions @ 60%-80% 1RM on the bench press, seated row, shoulder press, lat pulldown, biceps curl, triceps extension, leg press, leg extension, leg curl, abdominal crunch/curl, back extension), and cardiovascular training (walking or cycling for 20 to 30 min training at 60% to 80% heart rate reserve [HRR]). Additionally, participants will be asked to accumulate 10,000 steps per day of brisk walking on non-training days (goal > 100 min./wk. of moderate to vigorous exercise). Training will be recorded on training logs and by using an iPhone, Fitbit or pedometer.

Participants will be given 1,400, 1,500 kcal/day or 1,600 kcal/day diets based on resting energy expenditure determination designed to promote a 400-500 kcal/d energy intake deficit following the American Heart Association (AHA) macronutrient distribution recommendations (55% CHO, 30% FAT, 15% PRO). A goal energy intake, weekly diet plan, examples, and a food substitution list will be provided. A phone app (e.g., MyFoodDiary) will be used to help participants monitor and adhere to energy intake goals. In our prior studies, this exercise and diet intervention has been shown to promote a 3-5 kg fat loss, 3-5% decrease in percent body fat, a maintenance in fat free mass and REE, and improved health outcomes.

Primary Endpoints: Differences in body weight, body fat mass (kg and %), and waist and hip circumference at weeks 6 and 12 compared to baseline.

Secondary Endpoints: Differences in resting energy expenditure, aerobic capacity, estimated 1RM, muscular endurance total work, training volume, energy and macronutrient intake, blood lipids, and HbA1c, IL6, CRPhs, TNFa, INF, Leptin, HbA1C, Insulin, Glucose, Comprehensive Clinical Panel (HDL, LDL, TG, BUN, CREAT, etc.), side effects, SF-36 quality of life at weeks 6 and 12 compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Has given voluntary, written, informed consent to participate in the study;
2. Healthy pre-menopausal females age 18 - 50 years;
3. Body mass index (BMI) between 25 - 35 kg/m2 and/or body fat >30%; preferred BMI between 25-32 kg/m2; mean BMI in each group has to be in the range of 25-29.9.
4. Free-living (living in a private home, alone or with family, and able to maintain their health and hygiene without assistance);
5. In generally good health; and,
6. Willing to maintain consistent sleep duration the evening before study visits.

Mean average BMI will be controlled during phone screening. Anyone with a BMI from 25-29.9 (assuming other inclusion criteria are met with no exclusion criteria) will be enrolled and a list of alternatives for borderline subjects will be kept (e.g. up to 32). A log of active participants will be kept so subjects above 30 will not be added unless the mean is within 25-29.9 range

Exclusion Criteria:

1. Are pregnant, breastfeeding, or wish to become pregnant during the study;
2. Plan major changes in lifestyle (i.e. diet, dieting, exercise level, travel) during the study;
3. Have a recent history (<3 months) of exercise training or weight loss (> 5%);
4. Have an orthopedic limitation that would prevent participation in a general fitness program;
5. Have uncontrolled heart disease, hypertension, diabetes, thyroid disease, cancer, neurological disease, or untreated psychotic or major depressive disorder;
6. Have taken weight loss dietary supplements or medications during the last 4-wks;
7. Have a history of chronic use of oral or injectable corticosteroids;
8. Have a history within previous 12 months of alcohol or substance abuse;
9. Are a heavy smoking (>1 pack/day within past 3 months);
10. Have a history of heavy caffeinated beverage consumption (>400mg caffeine/day) within past 2 weeks; or,
11. Have known allergy to any of the ingredients in the supplement product or placebo.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Body fat mass (in Kg) | 6 and 12 weeks
  Difference in body fat mass (kg) evaluated by DEXA between weeks 6 and 12 compared to baseline.
Body fat mass (in % of total body weight) | 6 and 12 weeks
  Difference in body fat mass (% of total body weight) evaluated by DEXA between weeks 6 and 12 compared to baseline

SECONDARY OUTCOMES:
Total body weight (Kg) | 6 and 12 weeks
  Difference in total body weight between weeks 6 and 12 weeks compared to baseline
Waist circumference (cm) | 6 and 12 weeks
  Difference in waist circumference between weeks 6 and 12 weeks compared to baseline
Hip circumference (cm) | 6 and 12 weeks
  Difference in hip circumference between weeks 6 and 12 weeks compared to baseline
Resting energy expenditure (Kcal/day) | 6 and 12 weeks
  Difference in resting energy expenditure between weeks 6 and 12 weeks compared to baseline
Maximum oxygen uptake (ml/kg/min) | 6 and 12 weeks
  Difference in aerobic capacity between weeks 6 and 12 weeks compared to baseline
Muscle strenght - 1 Repetition Maximum (Kg) | 6 and 12 weeks
  Difference in estimated 1RM between weeks 6 and 12 weeks compared to baseline
Muscle strenght - 1 Repetition Maximum (% of estimated) | 6 and 12 weeks
  Difference in estimated 1RM between weeks 6 and 12 weeks compared to baseline
Muscular endurance total work (Kg) | 6 and 12 weeks
  Difference in muscular endurance total work between weeks 6 and 12 weeks compared to baseline
Energy daily intake (Kcal/day) | 6 and 12 weeks
  Difference in energy and macronutrient intake between weeks 6 and 12 weeks compared to baseline
Blood HDL-cholesterol level (g/l) | 6 and 12 weeks
  Difference in blood HDL-cholesterol level between weeks 6 and 12 weeks compared to baseline
Blood LDL-cholesterol level (g/l) | 6 and 12 weeks
  Difference in blood LDL-cholesterol level between weeks 6 and 12 weeks compared to baseline
Blood total cholesterol level (g/l) | 6 and 12 weeks
  Difference in blood total cholesterol level between weeks 6 and 12 weeks compared to baseline
Blood TGL level (g/l) | 6 and 12 weeks
  Difference in blood TGL level between weeks 6 and 12 weeks compared to baseline
blood TNFa level (pg/ml) | 6 and 12 weeks
  Difference in blood TNFa level weeks 6 and 12 weeks compared to baseline
blood INF level (pg/ml) | 6 and 12 weeks
  Difference in blood INF level weeks 6 and 12 weeks compared to baseline
blood IL6 level (pg/ml) | 6 and 12 weeks
  Difference in blood IL6 level weeks 6 and 12 weeks compared to baseline
blood CRPhs level (pg/ml) | 6 and 12 weeks
  Difference in blood CRPhs level weeks 6 and 12 weeks compared to baseline
Blood insulin level (mUI/l) | 6 and 12 weeks
  Difference in blood insulin level between weeks 6 and 12 weeks compared to baseline
Blood glucose level (mmol/l) | 6 and 12 weeks
  Difference in blood glucose level between weeks 6 and 12 weeks compared to baseline
Blood leptin level (ng/ml) | 6 and 12 weeks
  Difference in blood leptin level between weeks 6 and 12 weeks compared to baseline
Blood HbA1C level (%) | 6 and 12 weeks
  Difference in blood HbA1C level between weeks 6 and 12 weeks compared to baseline
Blood Creatinine level (umol/l) | 6 and 12 weeks
  Difference in blood Creatinine level between weeks 6 and 12 weeks compared to baseline
Blood total protein level (mmol/l) | 6 and 12 weeks
  Difference in blood total protein level between weeks 6 and 12 weeks compared to baseline
Blood Urea/BUN ratio (mmol/l) | 6 and 12 weeks
  Difference in blood Urea/BUN ratio between weeks 6 and 12 weeks compared to baseline
Blood Uric acid level (umol/l) | 6 and 12 weeks
  Difference in blood uric acid level between weeks 6 and 12 weeks compared to baseline
Blood AST level (U/l) | 6 and 12 weeks
  Difference in blood AST level between weeks 6 and 12 weeks compared to baseline
Blood ALT level (U/l) | 6 and 12 weeks
  Difference in blood ALT level between weeks 6 and 12 weeks compared to baseline
Quality of life score (SF-36) | 6 and 12 weeks
  Difference in quality of life score between weeks 6 and 12 weeks compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Richard B. Kreider, Principal Investigator — Exercise & Sport Nutrition Lab - Texas A&M University
Locations (1):
- Exercise & Sport Nutrition Lab, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dickerson B, Maury J, Jenkins V, Nottingham K, Xing D, Gonzalez DE, Leonard M, Kendra J, Ko J, Yoo C, Johnson S, Pradelles R, Purpura M, Jager R, Sowinski R, Rasmussen CJ, Kreider RB. Effects of Supplementation with Microalgae Extract from Phaeodactylum tricornutum (Mi136) to Support Benefits from a Weight Management Intervention in Overweight Women. Nutrients. 2024 Mar 28;16(7):990. doi: 10.3390/nu16070990. PMID 38613023
- [Derived] Yang M, Xuan Z, Wang Q, Yan S, Zhou D, Naman CB, Zhang J, He S, Yan X, Cui W. Fucoxanthin has potential for therapeutic efficacy in neurodegenerative disorders by acting on multiple targets. Nutr Neurosci. 2022 Oct;25(10):2167-2180. doi: 10.1080/1028415X.2021.1926140. Epub 2021 May 15. PMID 33993853